CLINICAL TRIAL: NCT06743906
Title: Role of OCT & OCT Angiography in Patients With Posterior at the Uveitis Clinic of Assiut University Hospital.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Lotfy Mahmoud Mohamed, resident doctor at Assiut University hospital, Assiut University
Other Study IDs: OCT & OCT posterior uveitis
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-04-21 (Actual); Status verified 2024-12

CONDITIONS: Uveitis, Posterior
Keywords: OCT & OCT angiography
MeSH Terms: conditions — Uveitis, Posterior; Ornithine Carbamoyltransferase Deficiency Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- uveitis patient: participants will be recruited from the ophthalmology outpatient clinic of Assiut University Hospitals.- Patient with posterior uveitis (infectious or non-infectious posterior uveitis).

SUMMARY:
OCT angiography is a recent evaluation of OCT technology which combines the structural assessment of ocular tissues obtained by OCT image with visualization of blood flow within the vessels in imaged area. So combined structural and function image can be obtained by OCT angiography.

Defferent type of uveitis often have specific OCT & OCT angiography findingwhich deffer according to the involved ocular tissue and according to the type of inflammatory / infectious process that characterize them.

The aim of study is to determine the role of OCT & OCT angiography in assessment of retinal and choroidal architectural and vascular changes in patients with posterior uveitis.

DETAILED DESCRIPTION:
Uveitis is a challenging disease. It represents a major cause of ocular morbidity worldwide. More than half of all patients with uveitis develop sight threatening complications related to their disease, and up to 35% of patients suffer severe visual impairment.

Uveitis and its complications are responsible for 5% to 10% of all causes of legal blindness in developed countries .

The causes of uveitis are numerous, and include infectious conditions, autoimmune diseases, trauma and tumors (masquerade syndrome). To develop an accurate differential diagnosis, clinicians must consider all available information, including the patient history, anatomic location of the inflammation (anterior or posterior), character (granulomatous vs. non granulomatous), laterality, and chronicity of inflammation. Moreover, diagnostic tools, such as fluorescein angiography (FA), indocyanine green angiography (ICG), optical coherence tomography (OCT) and ultrasound, play an important role in the diagnosis and in the management of the uveitis.

OCT & OCT angiography are now proven to be an effective noninvasive method in detecting pathologic features in uveitis and are rapidly gaining popularity as an ancillary exam. It may be used to assist in the diagnosis of uveitis and may be repeated safely during follow-up to monitor response to any intervention.

OCT angiography is a recent evaluation of OCT technology which combines the structural assessment of ocular tissues obtained by OCT image with visualization of blood flow within the vessels in imaged area. So combined structural and function image can be obtained by OCT angiography.

Defferent type of uveitis often have specific OCT & OCT angiography findingwhich deffer according to the involved ocular tissue and according to the type of inflammatory / infectious process that characterize them.

ELIGIBILITY:
Inclusion Criteria:

* - Patient age of greater than 18 years old.
* Patient can offer viable consent.
* Patient with posterior uveitis (infectious or non-infectious posterior uveitis).

Exclusion Criteria:

* - Patient unable to offer viable consent.
* Patient unwilling to participate.
* Any coexistence retinal pathology: diabetic retinopathy, other causes of retinal vascular occlusion, traumatic retinopathy, traumatic maculopathy, other peripheral ischemic retinopathy e.g. sickles cell retinopathy.
* Presence of media opacity hindering appropriate scan.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: participants will be recruited from the ophthalmology outpatient clinic of Assiut University Hospitals.- Patient with posterior uveitis (infectious or non-infectious posterior uveitis).
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
the choroidal thickness (CT) measurements | baseline
  The choroidal thickness (CT) measurements will be obtained from manual segmentation of OCT B-scans at the fovea for case numbers 1, 2, 4 and 5 and at the location of the choroiditis lesion

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gupta V, Gupta P, Singh R, Dogra MR, Gupta A. Spectral-domain Cirrus high-definition optical coherence tomography is better than time-domain Stratus optical coherence tomography for evaluation of macular pathologic features in uveitis. Am J Ophthalmol. 2008 Jun;145(6):1018-1022. doi: 10.1016/j.ajo.2008.01.021. Epub 2008 Mar 17. PMID 18343349
- [Background] Diniz B, Regatieri C, Andrade R, Maia A. Evaluation of spectral domain and time domain optical coherence tomography findings in toxoplasmic retinochoroiditis. Clin Ophthalmol. 2011;5:645-50. doi: 10.2147/OPTH.S20033. Epub 2011 May 17. PMID 21629569